CLINICAL TRIAL: NCT02488460
Title: Effects of a School-based Physical Activity Intervention on Math Achievement - A Randomized Controlled Trial
Brief Title: Effects of Physical Activity on Math - an RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: IMK Fonden (Other)
Responsible Party: Principal Investigator, Mona Have, PhD Fellow, Department of Sports Science and Clinical Biomechanics, University of Southern Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: h5vadgyk
Record Dates: First submitted 2015-06-08; First posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Academic Acheivement; Physical Activity
Keywords: Motor Activity; Cognition; Academic Acheivement; Preadolescent Children
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal math (No Intervention): This arm serves as the control group receiving regular math lessons
- Active math (Experimental): This arm serves as the intervention group receiving physically active math lessons
  Interventions: Behavioral: Physically active math lessons

INTERVENTIONS:
Behavioral: Physically active math lessons — The intervention consists of a nine month period with physical activity as part of, and integrated, in math lessons
  Arms: Active math

SUMMARY:
Background

Increased physical activity can improve cognition and academic skills. However due to economic concerns and increasing focus on standardized testing, PA in schools often receives little attention and physical education is reduced in many countries in favor of spending more time devoted to academic classes. This tendency is not compatible with the increasing evidence for the association between physical activity, fitness, cognitive and academic performance.

Despite increasing evidence for the association between PA, fitness, cognitive and academic performance, very few longitudinal high-quality studies exists examining the effect of physical activity on academic performance (ref.). Furthermore, to the best of our knowledge only two studies have assessed academic outcomes following the integration of physical activity into the classroom with intervention participants scoring significantly higher in test sections compared to controls which makes generalizing from these results challenging.

To promote policy changes that require more physical activity in school, empirical data are needed to study the effects of school-based physical activity programs. Therefore the investigators carried out a cluster randomized controlled trial conducted to examine the effect on math achievement and executive functions of classroom based PA in math.

DETAILED DESCRIPTION:
Study Design

Twelve elementary schools were cluster randomized to the active math intervention or served as control. Randomization was performed by shuffling sealed envelopes with intervention allocation inside to determine group assignment. This happened in a meeting where the leaders of the schools, employees at the municipalities and the responsible researcher were present. The study lasted for a school year (43 weeks) and the subjects were tested before and after the nine-month long intervention.

All tests were performed within one week except for the objective measurement of physical activity (PA) via accelerometer (ActiGraph, 7163, Pensacola, FL), which took place in a separate week, just before baseline and endline. In the intervention period (38 weeks) the participants received on average 6 mathematics lessons of 45 minutes per week with respectively physically active and traditional teaching.

The intervention

The intervention consisted of math teaching focusing on implementing PA in the classroom as a facilitating instrument. Teachers were told to include at least 15 minutes of physical activity in each 45 minutes math lesson. In addition sedentary activities were only allowed to last for maximum 20 minutes. Classroom-based PA had the aim of creating a meaningful binding between the mathematical concepts and a specific physical activity to improve mental representation of mathematics and thus contribute to understanding and memory of the mathematical concepts.

Classroom teacher training for implementation of the intervention

Training was provided to math teachers at each intervention school in a course given by the responsible group of researchers. The training was planned in collaboration between mathematics teachers in the intervention schools and the responsible group of researchers and was based on the curriculum for mathematics in Danish public schools. The planning of the teaching content took place on a 4-day mandatory course for all mathematics teachers with the purpose to enable the teachers to teach active mathematics and thereby to promote the math achievement.

As part of the course the teachers received a folder with suggestions for PA in math made by the responsible group of researchers. In addition they developed activities with specific instructions and inspiration for how teachers could incorporate PA as an element of academic instruction. Since the teacher's motivation and involvement can influence the outcome of the study, emphasis was placed on creating high motivation in the course by increasing understanding of the numerous positive cognitive effects of PA.

ELIGIBILITY:
Inclusion Criteria:

* 1st Grade primary school children on public schools

Exclusion Criteria:

* Physical disabilities
* No written informed consent from parents

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 545 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Math Skills, as measured by a 45-minute standardized math test specifically designed for this age group by the developer of the Danish national tests (MG) (Hoegrefe Forlag). | Change from Baseline Math Skills at 9 months
  During the first three weeks prior to randomization and intervention, and the last two weeks of the protocol after the intervention period.

SECONDARY OUTCOMES:
Cardiovascular Fitness, as measured by intermittent shuttle-run test (the Andersen intermittent running test). | Change from Baseline Cardiovascular Fitness at 9 months
  During the first three weeks prior to randomization and intervention, and the last two weeks of the protocol after the intervention period.
Body height as measured without shoes to the nearest 0.5 cm using Harpenden stadiometer (West Sussex, UK). Body mass as measured in light clothing to the nearest 0.1 kg using an electronic scale (Tanita BWB-800, Tokyo, Japan). | Change from Baseline Body Composition at 9 months
  During the first three weeks prior to randomization and intervention, and the last two weeks of the protocol after the intervention period.
Activity Behavior as measured by questionnaires sent via SMS | Short Message Service from the parents of the participant during the nine month long intervention period
  Once a week during the 9 month long intervention, the parents answered questions concerning the children's PA in leisure time and transportation to school.
Objective Physical Activity level, as measured by using accelerometry (ActiGraph, GT3X and GT3X+) | Change from Baseline Objective Physical Activity level at 9 months
  During the first three weeks prior to randomization and intervention, and the last two weeks of the protocol after the intervention period.
Physical Activity during Math Lessons, as measured by using accelerometry (ActiGraph, GT3X and GT3X+) | Change from Baseline Objective Physical Activity level during math lessons at 9 months
  During the first three weeks prior to randomization and intervention, and the last two weeks of the protocol after the intervention period.
Executive Functions, as measured by a modified Eriksen flanker task | Change from Baseline Executive Functions at 9 months
  During the first three weeks prior to randomization and intervention, and the last two weeks of the protocol after the intervention period.
Creativity, as measured by the Torrance Test of Creativity | Change from Baseline Creativity at 9 months
  During the first three weeks prior to randomization and intervention, and the last two weeks of the protocol after the intervention period.
Teacher Motivation, as measured by Short Message Service | Short Message Service during the last 6 months of the intervention period
  Once every month the teacher answers how motivated they feel to integrate PA in to the Math lessons
Excutive function, as measured by the BRIEF-questionnaire | Change from Baseline Executive Functions at 9 months
  During the first three weeks prior to randomization and intervention, and the last two weeks of the protocol after the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Mona H. Sørensen, PhD Fellow, Principal Investigator — University of Southern Denmark

REFERENCES:
- [Derived] Siersbaek GM, Have M, Wedderkopp N. The Effect of Leisure Time Sport on Executive Functions in Danish 1st Grade Children. Children (Basel). 2022 Sep 23;9(10):1458. doi: 10.3390/children9101458. PMID 36291397
- [Derived] Have M, Nielsen JH, Gejl AK, Thomsen Ernst M, Fredens K, Stockel JT, Wedderkopp N, Domazet SL, Gudex C, Grontved A, Kristensen PL. Rationale and design of a randomized controlled trial examining the effect of classroom-based physical activity on math achievement. BMC Public Health. 2016 Apr 11;16:304. doi: 10.1186/s12889-016-2971-7. PMID 27068574